CLINICAL TRIAL: NCT04780009
Title: Loupe-Based Intraoperative Fluorescence Imaging for the Guidance of Brain Tumor Surgery
Brief Title: Loupe-Based Intraoperative Fluorescence Imaging
Status: Recruiting | Type: Observational
Sponsor: Guoqiang Yu (Other)
Collaborators: Bioptics Technology LLC (Unknown); National Cancer Institute (NCI) (NIH); Kentucky Small Business Innovation Research / Small Business Technology Transfer (SBIR/STTR) (Unknown)
Responsible Party: Sponsor-Investigator, Guoqiang Yu, Professor, University of Kentucky
Organization: University of Kentucky (Other)
Other Study IDs: MCC-17-0605-F1V; R41CA243600-01 (NIH)
Record Dates: First submitted 2021-02-26; First posted 2021-03-03 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma Multiforme; Anaplastic Astrocytoma
Keywords: fluorescence; resection; 5-ALA; fluorescein; optical
MeSH Terms: conditions — Glioblastoma; Astrocytoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsies in and adjacent to the tumor will be collected for histopathology.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Glioblastoma multiforme (GBM) and anaplastic astrocytoma (AA) are the most common primary malignant brain tumors. Survival of patients with these brain tumors is directly related to the extent of resection. Consequently, a great deal of effort has been directed at developing techniques and technologies that allow more extensive, safe resections.

This study will test a loupe-based wearable device in the clinical setting and compare its accuracy with a large operative microscope to identify tumor tissues. Postoperative histopathological analysis on tumor tissues will be used as gold standards for comparison. The outcome from this study will be a low-cost, miniaturized, easy-to-operate, loupe-based fluorescence imaging device for intraoperative guidance of brain tumor resection with the same level of accuracy as the large microscope.

DETAILED DESCRIPTION:
This is a prospective, observational study to compare the measurement accuracies of a wearable loupe-based device and the large microscope against the gold standards of postoperative histopathological analysis on tumor tissues.

At the induction of anesthesia, patients will receive 5 mg/kg of intravenous sodium 5-aminolevulinic acid (5-ALA) or fluorescein. Surgery will be performed under the guidance of the operative fluorescence microscope (PENTERO with fluorescence kit + YELLOW 560, Carl Zeiss) or (PENTERO 900 + BLUE 400, Carl Zeiss). The operating room light will be dimmed for optimum reproduction of the fluorescent light. Tumor removal will be continued until no fluorescent area is visualized. To evaluate the accuracy of the device in the identification of tumor tissue, six samples will be biopsied from the tumor resection margin for each patient; three in the fluorescent area and three in the non-fluorescent area for the assessment of positive and negative predictive values of the devices, respectively. These biopsied tissues will be taken to the clinical pathology laboratory for the standard histological analysis.

To compare the accuracy of the two imaging systems in identifying tumor tissues, the tumor resection area will be visually observed by the surgeon and video recorded using the new loupe-based device at two time points (at least): immediately before and immediately after tumor removal. Additional fluorescence images may be taken during surgery as long as the surgical workflow is not impacted. Moreover, the four fresh biopsies (2 in the fluorescent area and 2 in the non-fluorescent area) taken from the tumor margin based on the operative microscope diagnosis will also be examined intraoperatively by the loupe-based device to determine whether they are fluorescent or non-fluorescent.

To discriminate between clear tumor tissue and the peritumoral areas, the postoperative histological analysis of the biopsied samples taken from the tumor margins will be classified on the basis of the current 2016 WHO classification. The neuropathologist will be blinded to the fluorescence characteristics of the biopsied samples.

ELIGIBILITY:
Inclusion Criteria:

* adults with brain malignant gliomas undergoing resection
* at least 18 years of age
* able to understand the consent

Exclusion Criteria:

* pregnant women
* under 18 years of age
* patients undergoing emergency surgery
* inability to give consent due to dysphagia or language barrier

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing glioblastoma multiforme and anaplastic astrocytoma resection recruited from the University of Kentucky Multidisciplinary Oncology Clinic (UK-MOC).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-11-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Positive Predictive Value (PPV) | 1 day
  The proportion of samples that are histologically confirmed as tumor-positive among all fluorescent samples will be calculated.
Negative Predictive Value (NPV) | 1 day
  The proportion of samples that are histologically confirmed as tumor-negative among all fluorescent samples will be calculated.

SECONDARY OUTCOMES:
Residual Tumor | 1 day
  The proportion of positive results among all tumors with residual as well as the proportion of negative results among tumors without residual will be calculated relative to post-operative histopathological analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Guoqiang Yu, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No